CLINICAL TRIAL: NCT06134765
Title: A Multi-cohort, Open-label, Multicenter Exploratory Clinical Study of Bemalenograstim Alfa for the Prevention of Reduced ANC in Patients With Colorectal Cancer/Pancreatic Cancer Following a Bi-weekly Chemotherapy
Brief Title: Bemalenograstim Alfa for the Prevention in Patients With Colorectal Cancer/Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0302
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bemalenograstim alfa for the prevention of reduced ANC in patients with colorectal/pancreatic cancer (Experimental): Patients with colorectal cancer and pancreatic cancer（N=32）receive FOLFOXIRI or mFOLFIRINOX with or without targeted therapy. Subcutaneous injection of Bemalenograstim alfa 20mg/ time 24-48h after each cycle of chemotherapy.
  Interventions: Drug: Bemalenograstim alfa
- Bemalenograstim alfa for the prevention of reduced ANC in patients with colorectal cancer (Experimental): Patients with colorectal cancer(N=57)receiving FOLFIRI with or without targeted therapy.Subcutaneous injection of Bemalenograstim alfa, 20mg/ time, 24-48h after each cycle of chemotherapy.
  Interventions: Drug: Bemalenograstim alfa

INTERVENTIONS:
Drug: Bemalenograstim alfa — Bemalenograstim alfa,20mg, once every treatment
  Other Names: F-627

SUMMARY:
A multi-cohort, open-label, multicenter exploratory clinical study of Bemalenograstim alfa for the prevention of reduced absolute neutrophil count(ANC) in patients with colorectal cancer/pancreatic cancer following a bi-weekly chemotherapy regimen.A total of 89 patients are planned to be enrolled.

DETAILED DESCRIPTION:
This multi-cohort, open-label, multicenter exploratory clinical study enrolled 89 patients with colorectal cancer and pancreatic cancer who were scheduled to receive at least 2 courses of a two-week chemotherapy regimen. The study was divided into two cohorts: Cohort 1 was colorectal cancer or pancreatic cancer patients receiving FOLFOXIRI or mFOLFIRINOX in combination with or without targeted drugs, and cohort 2 was colorectal cancer patients receiving FOLFIRI in combination with or without targeted drugs. Patients meeting the inclusion criteria received Bemalenograstim alfa injection (20mg/ time, subcutaneous injection) 24-48h after each course of chemotherapy, and Bemalenograstim alfa injection was used until the change of chemotherapy regimen or the fourth course of chemotherapy, whichever occurred first. After the subjects completed 2 courses of treatment, the follow-up treatment was carried out according to the diagnosis and treatment routine. Investigators need to ensure that the first course of chemotherapy is at the recommended dose; For the second to fourth course of treatment, delayed dosing or dose adjustment due to toxicity is allowed, and the chemotherapy dose is allowed to be adjusted by ±10%.

ELIGIBILITY:
Inclusion Criteria:

1. The patients voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up;
2. Age 18 and above, male or female;
3. Patients with locally advanced or advanced colorectal or pancreatic cancer confirmed by histology or cytology are scheduled to receive at least 2 courses of FOLFIRI, FOLFOXIRI, or mFOLFIRINOX with or without targeted therapy as part of first-line therapy (excluding those who relapse within 6 months after the end of adjuvant therapy) ;
4. Eastern Cancer Collaboration Group (ECOG) physical status (PS) score: 0-1;
5. Adequate organ and bone marrow function meets the following criteria:

   1. Blood routine examination standards should be met (no blood transfusion or blood products within 14 days, no G-CSF and other hematopoietic stimulating factors are used to correct): hemoglobin content (HB) ≥80g/L; Neutrophil count (ANC) ≥1.5×109/L; Platelet count (PLT) ≥100×109/L.
   2. Biochemical examination shall meet the following criteria: Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN); ALT and AST ≤ 2.5 ULN; If with liver metastasis, ALT and AST ≤ 5× ULN; Serum creatinine ≤ 1.5× ULN.
   3. Left ejection fraction >50%.
6. Infertile women, i.e. those who have been through menopause for at least one year or who have undergone sterilization (bilateral tubal ligation, double ovaries removal, or hysterectomy); Fertile patients agreed to use appropriate contraceptive methods: condoms, foam, gel, diaphragm, intrauterine device (IUD), birth control pills (given orally or by injection) for 1 month before the start of the trial and 30 days after the end of the study.
7. The investigators determined that the patient could tolerate the treatment of Bemalenograstim Alfa.

Exclusion Criteria:

1. Acute congestive heart failure, cardiomyopathy, or myocardial infarction as diagnosed by clinical, electrocardiogram or other means;
2. Rubber allergic people;
3. Patients who had received radiotherapy for bone lesions (patients who had received radiotherapy for lesions other than bone lesions could be enrolled 4 weeks later) ;
4. Have received a bone marrow or stem cell transplant;
5. Pregnant or lactating women;
6. Known to be seropositive for human immunodeficiency virus (HIV) or have AIDS;
7. Active tuberculosis disease; Or a recent history of contact with a person with TB, unless the tuberculin test is negative, Or tuberculosis patients undergoing treatment; Or a chest radiograph to check suspected cases;
8. Patients with alcohol or substance abuse, which affected their adherence to the study;以上
9. Known allergy to granulocyte colony-stimulating factors or excipients of drugs;
10. Received recombinant human granulocyte stimulating factor treatment within 6 weeks before inclusion;
11. Patients with a diagnosis of primary malignancy other than colorectal or pancreatic cancer were accompanied by the following, except: 1) malignancy in complete remission for at least 2 years prior to enrollment and without additional treatment during the study period; 2) non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence; 3) Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
12. Use of other investigational drugs within 1 month prior to study enrollment;
13. The investigators believe that the patients have diseases or symptoms that are not suitable for participation in the study and that the study drugs may harm the patient's health or affect the judgment of adverse events;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of reduced absolute neutrophil count(ANC) of grade ≥3 in the first cycle of chemotherapy | From Baseline to primary completion date, about 18 months
  The incidence of reduced absolute neutrophil count(ANC) of grade ≥3 in the first cycle of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, China